CLINICAL TRIAL: NCT05110118
Title: A Randomized, Double-blind, Single-dose, Parallel-group Study Comparing Pharmacokinetic Characteristics, Safety , Tolerability and Immunogenicity of LY01008 (Recombinant Humanized Anti-Human Vascular Endothelial Growth Factor Monoclonal Antibody Injection) and Avastin (Bevacizumab Injection) in Healthy Chinese Male Subjects
Brief Title: Pharmacokinetic Characteristics, Safety, Tolerability and Immunogenicity of LY01008 and Avastin in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY01008/CT-CHN-103
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer; Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Recurrent
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01008 (Experimental): Single intravenous injection of LY01008 3 mg/kg for 90 min(±1 min).
  Interventions: Drug: LY01008
- Avastin (Active Comparator): Single intravenous injection of Avastin 3 mg/kg for 90 min(±1 min).
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: LY01008 — Single intravenous injection
  Other Names: Recombinant Humanized Anti-Human Vascular Endothelial Growth Factor Monoclonal Antibody Injection
  Arms: LY01008
Drug: Avastin — Single intravenous injection
  Other Names: Bevacizumab
  Arms: Avastin

SUMMARY:
This is a randomized, double-blind, single-dose, parallel-group study comparing pharmacokinetic characteristics, safety , tolerability and immunogenicity of LY01008 (Recombinant Humanized Anti-Human Vascular Endothelial Growth Factor Monoclonal Antibody Injection) and Avastin (Bevacizumab Injection) in healthy Chinese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Subjects aged 18 - 45 years
* Subjects weighing ≥ 50.0 kg and ≤ 100.0 kg
* Subjects with a body mass index (BMI) ≥ 19.0 and ≤ 26.0 kg/m2

Exclusion Criteria:

* Subjects with evidence or history of clinically significant disease
* Subjects with a history of previous cancer
* Subjects with a history of hypertension, or abnormal blood pressure at screening/baseline measurements (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg confirmed by a repeat measurement on the same day)
* Subjects with a history of blood donation 3 months before study drug infusion
* Subjects with a history of exposure to antibodies 12 months before study drug infusion
* Subjects with previous exposure to anti-VEGF therapy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measurable concentration（AUC0-t） | From baseline to Day 99
Area under the plasma concentration-time curve from time zero to infinity（AUC0-∞） | From baseline to Day 99
Maximum (peak) plasma concentration（Cmax） | From baseline to Day 99
Chloride（CL） | From baseline to Day 99
Terminal elimination half-life（t1/2） | From baseline to Day 99
Apparent volume of distribution（Vd） | From baseline to Day 99

SECONDARY OUTCOMES:
Adverse Events(AEs) | From baseline to Day 99
Vital signs | From baseline to Day 99
Physical examinations | From baseline to Day 99
Clinical laboratory tests | From baseline to Day 99
12-lead ECGs | From baseline to Day 99
Positive rate of serum anti-drug antibody (ADA) | From baseline to Day 99
Positive rate of neutralizing antibody (NAb) | From baseline to Day 99

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou R, Yang J, Liu Y, Zhang Q, Lu C, Tang K, Li X, Tang W, Gao E, Wu C, Dou C, Hu W. A randomized, double-blind, parallel-group phase I study comparing the pharmacokinetics, safety, and immunogenicity of LY01008, a candidate bevacizumab biosimilar, with its reference product Avastin(R) in healthy Chinese male subjects. Expert Opin Biol Ther. 2022 Feb;22(2):263-269. doi: 10.1080/14712598.2022.2019703. Epub 2021 Dec 27. PMID 34913787